CLINICAL TRIAL: NCT02575222
Title: Phase I Study of Neoadjuvant Nivolumab in Patients With Non-metastatic High-risk Clear Cell Renal Cell Carcinoma
Brief Title: Study of Neoadjuvant Nivolumab in Patients With Non-metastatic Stage II-IV Clear Cell Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J15179; IRB00068726 (Other: JHMIRB)
Record Dates: First submitted 2015-10-06; First posted 2015-10-14 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: Immunotherapy; PD-1; anti-PD-1; antibody; Kidney Cancer; RCC; non-metastatic
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab (Experimental): 3 mg/kg, IV (in the vein) on day 1 of each 2-week cycle, for a total of 3 doses prior to nephrectomy.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — 3 mg/kg, IV (in the vein) on day 1 of each 2-week cycle, for a total of 3 doses prior to nephrectomy.
  Other Names: MDX-1106; BMS-936558; Opdivo

SUMMARY:
This study will evaluate the use of nivolumab before surgery in patients with high-risk clear cell renal cell carcinoma who are eligible for nephrectomy. Nivolumab is an antibody that may help activate the immune system by blocking the function of an inhibitory molecule, Programmed cell death-1 (PD-1).

ELIGIBILITY:
Inclusion Criteria (abbreviated):

1. Confirmed non-metastatic high-risk clear cell renal cell carcinoma (T2a-T4NanyM0 or TanyN1M0)
2. Schedule to undergo either partial or radical nephrectomy as part of treatment plan
3. Patient agrees to have a tumor biopsy
4. ECOG performance status of 0 or 1
5. Adequate organ and marrow function defined by study-specified laboratory tests
6. Must use acceptable form of birth control while on study and for approximately 31 weeks post-treatment completion
7. Willingness and ability to comply with scheduled visits, treatment plans, lab tests and other study procedures

Exclusion Criteria (abbreviated):

1. Other active malignancies within last 3 years (with some exceptions for skin, prostate, cervical, or breast cancer)
2. Need for urgent or emergent nephrectomy to relieve symptoms
3. Prior treatment for RCC including surgery, radiation, thermoablation or systemic therapy
4. Surgery within 28 days of starting study treatment (some exceptions for minor procedures)
5. Received live vaccine for infectious diseases within 28 days of starting study treatment
6. Prior treatment with any antibody or drug targeting T-cell costimulation or immune checkpoint pathways (anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, etc)
7. Use of immunosuppressive doses of systemic medications within 14 days prior to starting study drug.
8. Current use of immunosuppressive agents
9. History of severe hypersensitivity reaction to other monoclonal antibodies
10. Current signs or symptoms of severe progressive or uncontrolled hepatic, hematologic, gastrointestinal, endocrine, pulmonary or cardiac disease other than directly related to RCC
11. Uncontrolled psychiatric illness/social situations that would limit compliance with study requirements.
12. Active infection requiring therapy.
13. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
14. Positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA).
15. History of autoimmune disease or syndrome requiring systemic steroids or immunosuppressants (some exceptions apply).
16. Pulse oximetry of <92% on room air
17. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by number of participants experiencing adverse events | From the first dose of nivolumab treatment through 100 days post-surgery
  Number of participants experiencing any adverse event as defined by Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0)

SECONDARY OUTCOMES:
Objective Tumor Response Rate (by RECIST) | Assessed at baseline, prior to surgery, and 3 months after surgery
  Number of patients achieving a complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors (RECIST)
Objective Tumor Response Rate (by irRC) | Assessed at baseline, prior to surgery, and 3 months after surgery
  Number of patients achieving a complete response (CR) or partial response (PR) by immune-related response criteria (irRC)
Quality of Life as assessed by the Functional Assessment of Cancer Therapy-Kidney Symptom Index (FKSI) -15 questionnaire | Baseline, 2 weeks, 4 weeks, prior to surgery, and at 1-, 3-, 6-, and 12-months after surgery
  Total score range 0-60 with higher scores indicating a less symptomatic respondent.
Metastasis-Free Survival | 12 months post-operatively, then every 6 months for 5 years
  Number of months without evidence of metastasis.
Overall Survival | 12 months post-operatively, then every 6 months for 5 years
  Number of months alive.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad E Allaf, M.D, Principal Investigator — Department of Urology and The Brady Urological Institute at Johns Hopkins
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No